CLINICAL TRIAL: NCT07168980
Title: Intensive Chemotherapy Combined With Early, Adequate, and Intensive Use of Rituximab for Aggressive B-NHL in Children and Adolescents
Brief Title: Chemotherapy With Rituximab for Aggressive B-NHL in Children and Adolescents
Acronym: B-NHL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Nanjing Children's Hospital (Other); Children's Hospital of Soochow University (Other); West China Second University Hospital (Other); Qilu Hospital of Shandong University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Xiangya Hospital of Central South University (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-BNHL-2025
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mature B-cell Non-Hodgkin Lymphoma
Keywords: mature B-cell non-Hodgkin lymphoma; children; adolescent; rituximab
MeSH Terms: interventions — Cyclophosphamide; Vincristine; Cytarabine; Prednisone; Etoposide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Risk group 1 (Other): Complete resection of stage I or II disease: 3 courses (A-B-A) and 3 intrathecal injections(Cytarabine/Methotrexate/Dexamethasone, age adjusted);
  Interventions: Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone
- Risk group 2 (Other): Not or incompletely resected stage I/II disease and LDH <2ULN: 5 courses (A--B--A--B--A) and 8 intrathecal injections;
  Interventions: Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone
- Risk group 3 (Other): Stage III with LDH < 2 ULN, or Stage I,II with LDH in 2 to 4 ULN : Preface followed by 6 courses (P(Cyclophosphamide/Vincristine/Prednisone)-AA-BB-AA-BB-AA-BB) and 13 intrathecal injections(16 intrathecal injections with CNS2-3)
  Interventions: Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone; Drug: Prednisone,Vincristine, Cyclophosphamide
- Risk group 4 (Other): Stage III with LDH≥2ULN, or Stage IV, or B-AL: Preface followed by 6 dose of rituximab (375mg/m2) combined 6 courses of chemotherapy, together with 13 intrathecal injections((16 intrathecal injections with CNS2-3): P-(Rituximab-Rituximab)AA-(Rituximab-Rituximab)BB-(Rituximab)AA-(Rituximab)BB-AA-BB; stage IV or B-AL with LDH≥5ULN:P-(Rituximab-Rituximab)AA-(Rituximab-Rituximab)BB-(Rituximab)AA-(Rituximab)BB-AA-BB-AA-BB, together with 17 intrathecal injections((21 intrathecal injections with CNS2-3)
  Interventions: Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone; Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone; Drug: Prednisone,Vincristine, Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone — Cyclophosphamide 800mg/m2, D1, then 200mg/m2, D2~4;Vincristine 1.5mg/m2 (MAX 2mg), D1; Cytarabine 1g/m2/dose, (2 doses, 12-hour interval), D4; Doxorubincin 20mg/m2, D2,3; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1;
  Other Names: Protocol A
  Arms: Risk group 1
Drug: Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone — Ifosphamide 1.2g/m2, D1~5; Etoposide, 60mg/m2, D3~5; Methotrexate, 0.5g/m2, D1;Vincristine 1.5mg/m2 (MAX 2mg), D1; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1;
  Arms: Risk group 1
Drug: Cyclophosphamide, Vincristine, Cytarabine, Doxorubincin, Prednisone — Cyclophosphamide 800mg/m2, D1, then 200mg/m2, D2~4;Vincristine 1.5mg/m2 (MAX 2mg), D1; Cytarabine 1g/m2/dose, (2 doses, 12-hour interval), D4;Doxorubincin 20mg/m2, D2,3; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,8;
  Other Names: Protocol A
  Arms: Risk group 2
Drug: Ifosphamide, Etoposide, Methotrexate, Vincristine, Prednisone — Ifosphamide 1.2g/m2, D1~5; Etoposide, 60mg/m2, D3~5; Methotrexate, 0.5g/m2, D1;Vincristine 1.5mg/m2 (MAX 2mg), D1; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1
  Other Names: Protocol B
  Arms: Risk group 2
Drug: Cyclophosphamide, Vindelsine, Cytarabine, Doxorubincin, Prednisone — Cyclophosphamide 800mg/m2, D1, then 200mg/m2, D2~4; Vindelsine 3mg/m2 (MAX 5mg), D1; Cytarabine 2g/m2/dose, (2 doses, 12-hour interval), D4; Doxorubincin 20mg/m2, D2,3; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,4(CNS2-3),8
  Other Names: Protocol AA
  Arms: Risk group 3; Risk group 4
Drug: Ifosphamide, Etoposide, Methotrexate, Vindelsine, Prednisone — Ifosphamide 1.2g/m2, D1~5; Etoposide, 100mg/m2, D3~5; Methotrexate, 5g/m2, D1;Vindelsine 3mg/m2 (MAX 5mg), D1; Prednisone 60mg/m2, D1~7;Intrathecal injection, D1,8
  Other Names: Protocol BB
  Arms: Risk group 3; Risk group 4
Drug: Prednisone,Vincristine, Cyclophosphamide — Prednisone 45mg/m2, D1~7; Vincristine 1.5mg/m2(MAX 2mg), D1; Cyclophosphamide 300mg/m2, D1; Intrathecal injection, D1
  Arms: Risk group 3; Risk group 4

SUMMARY:
The purpose of this study is to test whether intensive chemotherapy combined with early, adequate, and intensive use of Rituximab for aggressive B-NHL in children and adolescents can improve the EFS and OS compared with the historical study CCCG-BNHL-2015.

DETAILED DESCRIPTION:
In our previous study (CCCG-BNHL-2015), four-year EFS was 88.3%, mostly owing to the use of Rituximab. However, four-year EFS was only 73% for group R4. And three-year EFS was even lower, 61% for stage IV and B-AL with LDH≥4ULN. To improve survival for pediatric patients with high risk B-NHL, the investigators launched a new study in China. In this study (CCCG-BNHL-2025), patients with stage III and LDH≥2ULN, any stage IV, and B-AL will be stratified into group R4. Six injections of Rituximab will be used for patients in R4, compared with four injections in CCCG-BNHL-2015. And two injections of Rituximab will be used in the first and second cycles of chemotherapies. The first cycle of chemotherapy will be changed into AA, instead of A. For patients with stage IV (including B-AL) with LDH≥ 4ULN, two cycles of chemotherapies(AA and BB) will be added. Our aim is to test whether intensive chemotherapies with early, adequate, and intensive use of Rituximab will improve the EFS and OS of children and adolescents with highly aggressive B-NHL.

ELIGIBILITY:
Inclusion Criteria:

Histology or cytologically confirmed matureB-cell NHL/AL(Burkitt, DLBCL, PMLBL,or aggressive mature B-cell NHL non other specified or specifiable) Able to comply with scheduled follow-up and with management of toxicity Signed informed consent

Exclusion Criteria:

Follicular lymphoma, MALT and nodular marginal zone are not included into this therapeutic study Patients with congenital immunodeficiency, chromosomal breakage syndrome, prior organ transplantation, previous malignancy of any type, or known positive HIV serology.

Evidence of pregnancy or lactation period. Past or current anti-cancer treatment except corticosteroids during less than one week.

Exclusion criteria related to rituximab:

Tumor cell negative for CD20. Prior exposure to rituximab. Hepatitis B carrier status history of HBV or positive serology.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi-jin Gao, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dong J, Xu Z, Guo X, Ye F, Fan C, Gao J, Gao Y, Yang L. Effect of rituximab on immune status in children with aggressive mature B-cell lymphoma/leukemia-a prospective study from CCCG-BNHL-2015. Heliyon. 2024 Mar 5;10(5):e27305. doi: 10.1016/j.heliyon.2024.e27305. eCollection 2024 Mar 15. PMID 38495131
- [Background] Zhao J, Liu TF, Wu KF, Yang LC, Xu XJ, Lu J, Shao JB, Li F, Ma FT, Guo X, Li H, Liu AG, Wang NL, Shen HP, Li Y, Liu SX, Liang CD, Shen SH, Fang YJ, Gao YJ. Clinical and molecular characteristics of paediatric mature B-cell acute lymphocytic leukaemia and non-Hodgkin lymphoma with bone marrow involvement: A joint study between the CCCG leukaemia and lymphoma groups. Br J Haematol. 2025 Apr;206(4):1149-1159. doi: 10.1111/bjh.20011. Epub 2025 Feb 17. PMID 39962993
- [Background] Wang X, Ding L, Fang Y, Yan J, Gao J, Yang L, Liu A, Lu J, Wang J, Zhang A, Gao Y, Ju X. The Prognostic and Risk Factors for Children With High-Risk Mature B-Cell Non-Hodgkin's Lymphoma: A Retrospective Multicenter Study. Cancer Med. 2024 Nov;13(21):e70309. doi: 10.1002/cam4.70309. PMID 39513286
- [Background] Minard-Colin V, Auperin A, Pillon M, Burke GAA, Barkauskas DA, Wheatley K, Delgado RF, Alexander S, Uyttebroeck A, Bollard CM, Zsiros J, Csoka M, Kazanowska B, Chiang AK, Miles RR, Wotherspoon A, Adamson PC, Vassal G, Patte C, Gross TG; European Intergroup for Childhood Non-Hodgkin Lymphoma; Children's Oncology Group. Rituximab for High-Risk, Mature B-Cell Non-Hodgkin's Lymphoma in Children. N Engl J Med. 2020 Jun 4;382(23):2207-2219. doi: 10.1056/NEJMoa1915315. PMID 32492302
- [Background] Gao YJ, Fang YJ, Gao J, Yan J, Yang LC, Liu AG, Ju XL, Lu J, Han YL, Wang J, Xie M, Guo X, Tang JY. A prospective multicenter study investigating rituximab combined with intensive chemotherapy in newly diagnosed pediatric patients with aggressive mature B cell non-Hodgkin lymphoma (CCCG-BNHL-2015): a report from the Chinese Children's Cancer Group. Ann Hematol. 2022 Sep;101(9):2035-2043. doi: 10.1007/s00277-022-04904-w. Epub 2022 Jul 13. PMID 35829780